CLINICAL TRIAL: NCT06259396
Title: The 8x5 Diet for Bile Acid Diarrhoea: A Feasibility Randomised Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Yvonne McKenzie, PhD Candidate, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19094
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Bile Acid Diarrhea
Keywords: diet intervention; nutrition; feasibility; diarrhoea; adults
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: feasibility randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The 8x5 Diet (Active Comparator): The 8x5 Diet is a healthy dietary pattern administered virtually by a specialist dietitian
  Interventions: Behavioral: The 8x5 Diet
- Control (No Intervention): Continuation of habitual diet, no dietary changes.

INTERVENTIONS:
Behavioral: The 8x5 Diet — A virtual, dietitian-counselled, healthy dietary pattern defined by its fat intake, its daily eating pattern, keeping adequately hydrated, having a variety of whole grains, fruit and vegetables, and use of certain plant fibres.
  Arms: The 8x5 Diet

SUMMARY:
Bile acid diarrhoea is a common cause of chronic watery diarrhoea. Treatment is life-long medication. However, about 50% of people have ongoing, bothersome diarrhoea. Findings from recent research on diet therapies and food intolerances have been used to develop a healthy dietary pattern called The 8x5 Diet. We will test the practicalities of conducting a randomised controlled trial of this dietary intervention.

DETAILED DESCRIPTION:
Bile acid diarrhoea is a lifelong gastrointestinal disorder that causes non-bloody and often urgent, diarrhoea. It is estimated that 1 in 100 adults in the United Kingdom are affected. To manage the diarrhoeal symptoms, daily oral medication is prescribed. About 50% of people are unable to achieve satisfactory symptom control, therefore other therapeutic options are needed. Recent research found a very high prevalence of perceived food intolerances with many people consequently avoiding foods. Systematic review of diet studies in bile acid diarrhoea showed that fat intake reductions and carbohydrate modification may have a beneficial effect on diarrhoea. However, no studies have been conducted as randomised controlled trials, undertaken outside of a hospital recruitment setting, or have assessed nutritional intakes and diet quality. With this paucity of evidence, The 8x5 Diet has been developed.

This study will be conducted virtually to recruit 76 adults from across the United Kingdom who are living with bile acid diarrhoea, have ongoing diarrhoea, and are without any other serious illnesses. Participants will be randomly allocated for 8 weeks to either their usual diet or to trial The 8x5 Diet with detailed advice from a specialist dietitian. The primary objective is to test the feasibility of the trial relating to consent, recruitment, randomisation, and retention. The results will inform the design of a future, definitive, and larger randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, of any ethnic group, living in the United Kingdom and not planning to move home for the next three months
* Self-reported diagnosis of bile acid diarrhoea that was confirmed by 7-day SeHCAT testing
* Self-reported ongoing chronic diarrhoea despite use of appropriate medication
* Able to participate in either diet group with the intention to remain in the group to which they were assigned for the 8 week study period
* Body mass index ≥20 kg m-2
* Able to converse in English (or via their carer, without assistance from an interpreter) using a computer/laptop, smart phone, or tablet
* Able to provide informed written consent
* Able to provide the address of their general practioner so that the research team can inform them of their participation.

Exclusion Criteria:

* Unable to provide self-reported written confirmation that their diagnosis of bile acid diarrhoea was by SeHCAT testing
* Pregnant/breastfeeding/planning a pregnancy in the next six months
* Inflammatory bowel disease, previous or current microscopic colitis, or other serious morbidities such as liver disease, pancreatic disease, AIDS/HIV, radiotherapy for cancer, assessed at screening via patient self-report
* Diarrhoea that is inadequately active: <3 stools per day or <1 watery stool (Bristol Stool Form types 6-7) per day as the mean of one week
* Currently participating in another research study or has taken part in the previous 3 months
* If taking insulin, metformin (other than slow-release), anti-obesity medication, or using commercially available formulated supplements to replace meals in previous three months
* Use of antibiotics in the previous four weeks

Medically necessary dietary exclusions or issues deemed incompatible with the trial:

* Food allergies, other than oral allergy syndrome/pollen-food syndrome
* Exclusion of gluten (i.e. coeliac disease), lactose, biogenic amines, or any other dietary exclusion assessed as unsuitable as screening by the trial team. This includes if the participant knows they would refuse to eat: starchy foods, fruit and vegetables, protein-rich foods, or dairy and alternatives (e.g. following a ketogenic diet)
* An eating disorder or disordered eating which is active or in the last 12 months
* Alcohol or drug abuse, or self-harm, or depression, or suicide ideation in the last 12 months
* Shift worker
* If unwilling to keep a weighed 7-day food diary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Consent | Recruitment period (50 weeks)
  The number (%) of participants who consent to participate in the trial compared to the number (%) that were screened by the research team.
Recruitment | Recruitment period (50 weeks)
  The number (%) of participants randomised compared to the number (%) that were eligible (screened by the research team)
Randomisation | Recruitment period (50 weeks)
  The number (%) of participants who complete their first appointment compared to the number (%) that were randomised, intervention group only.
Retention | Randomisation to trial completion (8 weeks)
  Tthe number (%) of participants that completed the study compared to the number (%) randomised to each group.
The trial's data collection instruments and procedures: Missing data | At baseline and at Week 8
  The number and proportion of missing data identified by the research team from questionnaires.
The trial's data collection instruments and procedures: Participants' views and experiences | Study identification to study completion (Week 8)
  Participants' views and experiences of the instruments (questionnaires and diaries) and procedures (screening, randomisation, baseline period, trial, general)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Todd, Professor, Study Chair — The University of Manchester
Locations (1):
- Yvonne McKenzie, Manchester, Greater Manchester, United Kingdom

REFERENCES:
- [Derived] McKenzie YA, Kelman L, O'Connor M, Todd C, Walters JR, Burden S. Diet therapy (The 8x5 Diet) for adults living with bile acid diarrhoea: protocol for a feasibility randomised controlled trial. BMJ Open. 2025 Mar 27;15(3):e097973. doi: 10.1136/bmjopen-2024-097973. PMID 40147991